CLINICAL TRIAL: NCT07275320
Title: Comparison of the Effects of Ultrasound-Guided Cervical Retrolaminar Block and Fluoroscopy-Guided Cervical Epidural Injection in Cervical Radiculopathy
Brief Title: Cervical Retrolaminar Block Versus Cervical Epidural Injection for Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Natia Arveladze, Anesthesiologist, Department of Anesthesiology and Reanimation, Istanbul Medeniyet University; Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRLB-ANEST-NA-O1
Record Dates: First submitted 2025-11-17; First posted 2025-12-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical retrolaminar block; Cervical epidural steroid injection; Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: This study was conducted using a parallel assignment design. A total of 70 patients with cervical radiculopathy unresponsive to conservative management were randomized in a 1:1 ratio to two groups using a sealed-envelope method. Group 1 was assigned to receive fluoroscopy-guided cervical epidural injection (ESI), and Group 2 was assigned to receive ultrasound-guided cervical retrolaminar block (CRLB). All participants were prospectively followed for 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: The clinician responsible for follow-up visits and outcome assessments (VAS and NDI) was blinded to the type of block performed in order to ensure objective evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRUP 1: Fluoroscopy-guided cervical interlaminar epidural Injection (Active Comparator): Participants in Group 1 are treated with a fluoroscopy-guided cervical interlaminar epidural injection consisting of 8 mL of a solution containing 0.25% bupivacaine and 8 mg dexamethasone.
  Interventions: Procedure: Fluoroscopy-guided cervical interlaminar epidural injection; Drug: Bupivacaine 0.25%; Drug: Dexamethasone
- Group 2 - Ultrasound-guided cervical retrolaminar block (Active Comparator): Participants in Group 2 are treated with an ultrasound-guided cervical retrolaminar block using a solution containing 0.25% bupivacaine and 8 mg dexamethasone. The injectate is administered either unilaterally with 4 mL or bilaterally with a total of 8 mL, depending on the patient's symptoms.
  Interventions: Procedure: Cervical Retrolaminar Block; Drug: Bupivacaine 0.25%; Drug: Dexamethasone

INTERVENTIONS:
Procedure: Fluoroscopy-guided cervical interlaminar epidural injection — A fluoroscopy-guided cervical interlaminar epidural injection was performed as a non-surgical treatment option for cervical radiculopathy. Under C-arm fluoroscopic guidance, the C7-T1 intervertebral space was identified. An 18-gauge Tuohy needle was advanced into the epidural space via a medial approach using the hanging drop technique. After confirming epidural spread with the injection of 1 mL of non-ionic contrast solution, an epidural injection was performed with a total of 8 mL of solution containing 0.25% bupivacaine and 8 mg dexamethasone.
  Arms: GRUP 1: Fluoroscopy-guided cervical interlaminar epidural Injection
Procedure: Cervical Retrolaminar Block — patients who received a cervical retrolaminar block were administered a solution containing 0.25% bupivacaine and 8 mg dexamethasone under ultrasound guidance. The injectate was applied unilaterally with 4 mL or bilaterally with a total of 8 mL, depending on the patient's symptoms
  Arms: Group 2 - Ultrasound-guided cervical retrolaminar block
Drug: Bupivacaine 0.25% — Bupivacaine 0.25% solution is used as the local anesthetic component of both the fluoroscopy-guided cervical interlaminar epidural injection and the ultrasound-guided cervical retrolaminar block.
Drug: Dexamethasone — Dexamethasone 8 mg is used as the corticosteroid component of both the fluoroscopy-guided cervical interlaminar epidural injection and the ultrasound-guided cervical retrolaminar block.

SUMMARY:
Cervical radiculopathy is a common clinical condition, affecting approximately 1 in 1,000 individuals each year, and is typically characterized by neck pain radiating to the upper extremities. Although about 90% of patients respond to conservative treatment, cervical epidural steroid injection is widely used as an interventional alternative to surgery in those with symptoms refractory to conservative management. However, concerns regarding the safety of cervical epidural steroid injection have increased in recent years. Ultrasound-guided cervical retrolaminar block, which does not require entry into the neuraxial space, is considered a theoretically safer technique.

In this prospective, randomized study, 70 patients with cervical radiculopathy refractory to conservative treatment were enrolled and randomly assigned to receive either ultrasound-guided cervical retrolaminar block (n = 35) or fluoroscopy-guided cervical epidural steroid injection (n = 35). The study aimed to compare the clinical efficacy and safety of these two interventional approaches.

DETAILED DESCRIPTION:
Cervical radiculopathy is the fourth leading cause of disability in the United States. In the general population, the lifetime risk of developing neck pain is approximately 50%. Cervical radiculopathy is a common clinical condition, often presenting with neck pain radiating to the upper extremities, with an annual incidence of approximately 1.79 per 1,000 individuals. The natural course of cervical radiculopathy tends toward spontaneous recovery in more than 90% of patients. First-line treatment options are generally non-surgical and include analgesics, cervical stabilizing exercises, traction, and physical therapy. In patients requiring surgery, the most frequently applied procedures are decompression with or without fusion. However, cervical spine surgery carries important risks and complications. Reported complication rates include surgical site infection (0.7-4%), dysphagia in more than 20% of patients, nerve root injury in up to 12%, and spinal cord injury in approximately 0.01%. Cervical epidural steroid injection is one of the most widely used cervical interventions and provides a non-surgical alternative. In patients refractory to conservative treatment but without progressive neurological deficit, cervical epidural steroid injections are commonly recommended. Nevertheless, there is currently no consensus on the optimal technique that best balances safety and efficacy. In recent years, paraneuraxial interfascial blocks performed under ultrasound guidance have gained popularity due to their anatomical and clinical advantages. Cervical retrolaminar block belongs to this group. In this technique, the injectate is administered between the lamina of C6 or C7 and the multifidus muscle, where there are no critical vascular or neural structures; for example, the deep cervical artery courses more laterally. A more medial approach may also reduce the risk of phrenic nerve paresis. In contrast, cervical epidural injections are less localized and may be associated with systemic side effects such as hypotension, urinary retention, and motor impairment. Ultrasound-guided cervical retrolaminar block offers several potential advantages, including technical simplicity due to clear bony landmarks, a lower risk of vascular injury, a reduced likelihood of phrenic nerve involvement or systemic adverse effects, and avoidance of radiation exposure. The hypothesis of this study was that ultrasound-guided cervical retrolaminar block is non-inferior to fluoroscopy-guided cervical epidural steroid injection in terms of pain relief and functional improvement in patients with cervical radiculopathy refractory to conservative treatment, while potentially offering a safer alternative. This trial was conducted as a prospective, randomized, controlled study at Istanbul Medeniyet University, Faculty of Medicine, Goztepe Prof. Dr. Suleyman Yalcin City Hospital. Written informed consent was obtained from all participants prior to enrollment, and the study was performed in accordance with international ethical standards and the Declaration of Helsinki. A total of 70 patients were included. Eligible participants were between 18 and 80 years of age, had MRI-confirmed cervical radiculopathy with a clearly identified affected level, and presented with pain intensity of at least 5 on the Visual Analog Scale (VAS) and an elevated Neck Disability Index (NDI) score. Additional inclusion criteria were absence of motor weakness, absence of signs or symptoms of myelopathy, and refractoriness to conservative treatments including manipulation, traction, physical therapy, and oral analgesics. Exclusion criteria included refusal to provide consent; coagulopathy; allergy or intolerance to local anesthetics; severe organ failure; pregnancy or lactation; cervical spine or adjacent soft tissue infection; inflammatory rheumatologic disease; fibromyalgia; neurological or neuromuscular disorders; demyelinating diseases; polyneuropathy; congenital malformations; prior cervical spine surgery; and comorbidities such as carpal tunnel syndrome, cubital tunnel syndrome, thoracic outlet syndrome, brachial plexus injury, or shoulder pathology. Patients who had previously received local corticosteroid injections, those using neuropathic pain agents (e.g., pregabalin, gabapentin), and those with cardiac pacemakers were also excluded. Patients were randomized into two groups. Group 1 (n = 35) received interlaminar cervical epidural steroid injection under fluoroscopic guidance, and Group 2 (n = 35) underwent ultrasound-guided cervical retrolaminar block. Randomization was performed using a sealed-envelope method. Following group allocation, all patients were informed about the assigned procedure and signed a standardized written informed consent form that detailed the study objectives, duration, interventions, and potential risks. Patient assessments included baseline and post-procedural evaluations using the Visual Analog Scale and the Neck Disability Index. Measurements were recorded at baseline (VAS-0, NDI-0) and at weeks 1 (VAS-1, NDI-1), 4 (VAS-4, NDI-4), 8 (VAS-8, NDI-8), and 12 (VAS-12, NDI-12). Additional recorded variables included patient age, sex, side of block application, need for surgery during follow-up, and adverse effects or complications related to the procedures or local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cervical radiculopathy confirmed by magnetic resonance imaging (MRI).
* Visual Analog Scale (VAS) pain score ≥ 5 and an elevated Neck Disability Index (NDI) score.
* Age between 18 and 80 years.
* Patients without motor weakness or clinical signs of myelopathy.
* Patients who did not respond to conservative treatments such as analgesics, physical therapy, or traction.

Exclusion Criteria:

* Patients who do not provide informed consent or who have coagulopathy.
* Patients with a known allergy to the study medications, organ failure, pregnancy, or lactation.
* Patients with infection in the cervical spine or surrounding tissues, or those with rheumatologic, neurologic, or neuromuscular diseases.
* Patients with a history of cervical spine surgery or with shoulder/peripheral nerve pathology that may confound the diagnosis.
* Patients using neuropathic pain medications (such as pregabalin or gabapentin) or those with a cardiac pacemaker.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity assessed by the Visual Analog Scale (VAS) | At baseline and at 1, 4, 8, and 12 weeks after the procedure.
  Pain intensity will be assessed in both groups using a 10-cm Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain." VAS scores will be recorded before the procedure (baseline) and at 1, 4, 8, and 12 weeks after the intervention. The primary outcome is the change in VAS pain scores from baseline at 1, 4, 8, and 12 weeks and the comparison of these changes between the two treatment groups.

SECONDARY OUTCOMES:
Change in Neck Disability Index (NDI) score | At baseline and at 1, 4, 8, and 12 weeks after the procedure.
  Functional disability will be evaluated using the Neck Disability Index (NDI). NDI scores will be recorded in both groups before the procedure (baseline) and at 1, 4, 8, and 12 weeks after the intervention. The secondary outcome is the change in NDI score from baseline at 1, 4, 8, and 12 weeks and the comparison of these changes between the two treatment groups.
Incidence of treatment-related adverse events in both groups | Day of the procedure (baseline) to 12 weeks after the intervention
  All procedure-related adverse events were recorded in both groups from the day of the procedure to 12 weeks after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: MAHMUT DURMUS, Prof. Dr., MD, Study Chair — Department of Anesthesiology and Reanimation, Interventional Pain (Algology) Unit, Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Istanbul Medeniyet University
Locations (1):
- Goztepe Suleyman Yalcin City Hospital, Department of Anesthesiology and Reanimation, Interventional Pain Management Unit, Istanbul, Kadikoy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No